CLINICAL TRIAL: NCT00160498
Title: A Double-Blind, Randomized, Multicenter, Placebo-Controlled, Parallel, Dose-Titration Study to Assess the Efficacy of Lercanidipine 10 mg and 20 mg Once Daily p. o. in Hypertensive Subjects (I or II WHO) With Elevated Body Weight.
Brief Title: Testing the Efficacy of Different Dosages of Lercanidipine to Reduce Hypertensive Blood Pressure in Normal Weight and Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Ler 25-03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-03

CONDITIONS: Hypertension
Keywords: Lercanidipine, calcium antagonist, hypertension, obesity
MeSH Terms: conditions — Hypertension; Obesity | interventions — lercanidipine

INTERVENTIONS:
Drug: Lercanidipine

SUMMARY:
A double blind study to examine the safety and efficacy of different dosages of lercanidipine in normal weight and obese patients with hypertension

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): 18.0 - 24.9 or 30.0 - 39.9 kg/m2 (extremes included);
* Essential hypertension I or II WHO:
* 140 mmHg ≤ BPs ≤ 179 mmHg and BPd ≤ 109 mmHg at the end of the placebo run-in phase;

Exclusion Criteria:

* Secondary hypertension;
* Diabetes mellitus type 1, insulin dependent diabetes mellitus type 2, fasting blood glucose ≥ 160 mg/dl;
* Subjects keeping to a hypocaloric diet (except special diet for diabetics) to reduce body weight;
* History or presence of angioneurotic oedema;
* Subjects developing a hypertensive crisis during wash-out or placebo run-in period;

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2004-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
change from baseline of systolic blood pressure (BPs) after 4 weeks of treatment

SECONDARY OUTCOMES:
Blood pressure, response rate, normalization rate, pulse rate, lipid profile, safety and tolerability. Measures after 4, 8, 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Scholze, MD, Study Director — UCB Pharma